CLINICAL TRIAL: NCT02508194
Title: A Phase 2b Randomized, Double-blind Study to Evaluate the Efficacy of MEDI7510 for the Prevention of Acute Respiratory Syncytial Virus-associated Respiratory Illness in Older Adults
Brief Title: A Study to Evaluate the Efficacy of MEDI7510 in Older Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Year 1 of study completed. No enrollment planned for Year 2 of study.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D4420C00005
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Respiratory Syncytial Virus
Keywords: RSV; Older adults; MEDI7510; Vaccine; Efficacy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo + Inactivated Influenza Vaccine (IIV) (Active Comparator): Participants received a single intramuscular (IM) injection of placebo (matched with MEDI7510) in one arm and single IM injection of (IIV) in the contralateral arm.
  Interventions: Biological: IIV; Other: Placebo
- MEDI7510 + IIV (Experimental): Participants received a single IM injection of MEDI7510 in one arm and single IM injection of IIV in the contralateral arm.
  Interventions: Biological: MEDI7510; Biological: IIV

INTERVENTIONS:
Biological: MEDI7510 — RSV soluble fusion protein (sF) antigen plus glucopyranosyl lipid A in stable emulsion (GLA-SE) adjuvant
  Arms: MEDI7510 + IIV
Biological: IIV — Marketed Inactivated Influenza Vaccine
Other: Placebo — Sterile Saline
  Arms: Placebo + Inactivated Influenza Vaccine (IIV)

SUMMARY:
This study will be the first assessment of the efficacy of MEDI7510 for the prevention of respiratory syncytial virus (RSV) disease. It will also provide estimates of vaccine efficacy and of endpoint incidence in the placebo arm. It will also assess the safety and immunogenicity of concurrent dosing of MEDI7510 and IIV to expand on the observations made in the Phase 1b study of MEDI7510. It will also expand the safety database of participants dosed with MEDI7510. The study will also assess the immune response to MEDI7510 in Season 1 and Season 2.

DETAILED DESCRIPTION:
A Phase 2b, double-blind, randomized, and controlled study to evaluate the efficacy of MEDI7510 in approximately 1,900 adult participants, globally, 60 years or older. Participants will be randomized in a 1:1 ratio to receive a single intramuscular dose of each of 2 study vaccines in contralateral arms: MEDI7510 + IIV or placebo + IIV in Season 1.

Participants who receive MEDI7510 in the Northern Hemisphere will be re-randomized and blinded in Season 2 to receive either MEDI7510 + IIV or placebo + IIV in a 1:1 ratio. Clinical efficacy will not be assessed in Season 2; however the safety of revaccination will be assessed in Season 2.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years at the time of screening.
* Medically stable such that, according to the judgment of the investigator, hospitalization within the study period is not anticipated and the subject appears likely to be able to remain in follow-up through the end of protocol-specified follow-up.
* (Season 2): Subject received MEDI7510 and IIV in the Northern Hemisphere in Season 1.

Exclusion Criteria:

* History of allergy to any component of the vaccine.
* Receipt of seasonal influenza vaccine within 6 months prior to Season 1 dosing.
* History of allergy to or intolerance of IIV.
* Pregnancy or potential to become pregnant during the study. Females who (1) have had a menstrual period within the 12 months prior to study enrollment or (2) are undergoing any fertility treatment or who plan to undergo fertility treatments during the study period are excluded.
* History of Guillain-Barré syndrome.
* Previous vaccination against RSV.
* History of allergy to eggs in adulthood.
* History of or current autoimmune disorder, with the exception of stable, treated hypothyroidism caused by autoimmune thyroiditis, which is acceptable.
* Immunosuppression caused by disease, including human immunodeficiency virus infection (assessed by history), or medications. Any receipt of oral or intravenous glucocorticoid therapy within 30 days prior to enrollment or planned dosing within the follow-up period would disqualify. Topical, intranasal, inhaled, or intra-articular corticosteroids do not disqualify. Expected need for immunosuppressive medications during the follow-up period would disqualify.
* History of cancer within preceding 5 years other than treated non-melanoma skin cancer, locally-treated cervical cancer or in situ carcinoma of the breast.
* Receipt of any non-study vaccine within 28 days prior to study dosing or expected receipt of non-study vaccine prior to the Day 29 visit in Season 1.
* Receipt of any investigational product (IP) in the 90 days prior to randomization or expected receipt of IP during the period of study follow-up.
* Receipt of immunoglobulins or blood products within 4 months of study dosing (120 days) or expected receipt of immunoglobulins or blood products during the period of study follow-up.
* Current bleeding or clotting disorder including use of anticoagulants other than drugs with anti-platelet activity (such as nonsteroidal anti-inflammatory drugs, clopidogrel, ticagrelor or aspirin).
* History of alcohol or drug abuse or psychiatric disorder that, in the opinion of the investigator, would affect the subject's safety or compliance with study.
* (Season 2): Related Grade 3 or 4 adverse event (AE) including Grade 3 or 4 local reaction to either MEDI7510 or IIV, any adverse event of special interest (AESI) for an adjuvanted vaccine, or any related serious adverse event (SAE).

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1900 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2016-09-09 (Actual); Study Completion 2016-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (30):
  - Research Site, Sacramento, California
  - Research Site, San Francisco, California
  - Research Site, Aurora, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Lady Lake, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Savannah, Georgia
  - Research Site, Champaign, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Council Bluffs, Iowa
  - Research Site, Augusta, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Edina, Minnesota
  - Research Site, Cincinnati, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Bellevue, Nebraska
  - Research Site, Norfolk, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Rochester, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Dakota Dunes, South Dakota
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Murray, Utah
- Canada (5):
  - Research Site, Brampton, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Québec
- Chile (2):
  - Research Site, Santiago
  - Research Site, Temuco
- Estonia (2):
  - Research Site, Paide
  - Research Site, Tallinn
- Latvia (3):
  - Research Site, Daugavpils
  - Research Site, Jelgava
  - Research Site, Kuldīga
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- South Africa (7):
  - Research Site, Bellville
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Johannesburg
  - Research Site, Krugersdorp
  - Research Site, Pretoria
  - Research Site, Somerset West

REFERENCES:
- [Derived] Chang LA, Phung E, Crank MC, Morabito KM, Villafana T, Dubovsky F, Falloon J, Esser MT, Lin BC, Chen GL, Graham BS, Ruckwardt TJ. A prefusion-stabilized RSV F subunit vaccine elicits B cell responses with greater breadth and potency than a postfusion F vaccine. Sci Transl Med. 2022 Dec 21;14(676):eade0424. doi: 10.1126/scitranslmed.ade0424. Epub 2022 Dec 21. PMID 36542692
- [Derived] Falloon J, Yu J, Esser MT, Villafana T, Yu L, Dubovsky F, Takas T, Levin MJ, Falsey AR. An Adjuvanted, Postfusion F Protein-Based Vaccine Did Not Prevent Respiratory Syncytial Virus Illness in Older Adults. J Infect Dis. 2017 Dec 12;216(11):1362-1370. doi: 10.1093/infdis/jix503. PMID 29029260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1900 participants were randomized and participated in the study at 60 sites in 7 countries.
Pre-assignment Details: A total of 2,044 participants were screened, of which 144 participants were screen failures and 1900 participants were randomized in the study.
Period: Overall Study
Arm/Group | Placebo + Inactivated Influenza Vaccine (IIV) | MEDI7510 + IIV
Started | 949 | 951
Completed | 897 | 907
Not Completed | 52 | 44
Not completed — Death | 5 | 3
Not completed — Lost to Follow-up | 25 | 18
Not completed — Withdrawal by Subject | 20 | 18
Not completed — Error in Randomization | 1 | 3
Not completed — Principal Investigator Decision | 1 | 2

BASELINE CHARACTERISTICS:
Population: As-treated population (ATP): Participants who received any dose of investigational product (IP). Participants were included in the ATP according to the IP received even if different from that to which the participant was randomized.
Groups:
- Placebo + IIV: Participants received a single IM injection of placebo (matched with MEDI7510) in one arm and single IM injection of IIV in the contralateral arm.
- Total: Total of all reporting groups
Arm/Group | Placebo + IIV | MEDI7510 + IIV | Total
Number analyzed (Participants) | 949 | 951 | 1900
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.1 (6.2) | 68.1 (6.3) | 68.1 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 587 | 530 | 1117
  Male | 362 | 421 | 783

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had a First Episode of Acute Respiratory Syncytial Virus-Associated Respiratory Illness (ARA-RI) During Respiratory Syncytial Virus (RSV) Surveillance Period in Season 1
Description: ARA-RI was defined as an event in which a participant met specified clinical criteria and the event was laboratory-confirmed to be RSV-related. The specified clinical criteria included a minimum of 1 symptom from any 2 of the 3 symptom columns: one symptom from upper respiratory symptom column and one symptom from lower respiratory symptom column; one symptom from upper respiratory symptom column and one symptom from systemic symptom column; or one symptom from lower respiratory column and one from systemic symptom column and laboratory confirmation of RSV on at least 1 sample obtained between Day 1 to Day 8 of illness. The surveillance period was approximately 7 months and Season 1 was approximately 1 year.
Time Frame: Day 14 after dosing through end of surveillance period (approximately 7 months)
Population: Per-protocol population: All participants in the as-treated population (ATP) who were followed for qualifying symptoms for RSV until the end of the RSV surveillance period. Participants who met the primary endpoint criteria and were not followed until the end of the RSV surveillance period were also included in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 935 | 931
Percentage of Participants | 1.6 | 1.7
Statistical Analysis 1: Comparison: Placebo + IIV vs MEDI7510 + IIV; 2 sided 90 percent (%) confidence interval (CI) was used to compare vaccine efficacy (VE). VE = ([1 - relative risk (RR)] *100%), where RR was the RR of ARA-RI in the MEDI7510 group compared with the placebo group. A lower bound of the 90% CI greater than (>) 0% would demonstrate the efficacy of MEDI7510; Test type: Superiority; Vaccine efficacy = -7.1, 90% CI 2-sided [-106.9 to 44.3] — The CI was estimated by an exact conditional method

2. Secondary Outcome: Percentage of Participants Who Had a RSV Polymerase Chain Reaction (PCR)-Positive Respiratory Illness During the RSV Surveillance Period in Season 1
Description: Detection of RSV was done by PCR method by using any respiratory sample. The incidence of RSV PCR-positive respiratory illness during the RSV surveillance period was evaluated. The surveillance period was approximately 7 months and Season 1 was approximately 1 year.
Time Frame: Day 14 after dosing through end of surveillance period (approximately 7 months)
Population: Per-protocol population: All participants in the ATP who were followed for qualifying symptoms for RSV until the end of the RSV surveillance period. Participants who met the primary endpoint criteria and were not followed until the end of the RSV surveillance period were also included in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 935 | 931
Percentage of Participants | 1.6 | 1.7

3. Secondary Outcome: Geometric Mean Responses (GMRs) of Serum Antibodies Concentration Against RSV by Anti-Fusion Protein (F) Immunoglobulin G (IgG) Assay
Description: Anti-F IgG antibodies concentration were determined by a multiplex IgG assay developed on the Meso Scale discovery platform. It was calculated as: anti-log2 [mean (log2 xi)], where "xi" is an antibodies concentration of participants. The Season 1 was approximately 1 year.
Time Frame: Day 1, Day 29, and End of Season 1 (approximately 1 year)
Population: Immunogenicity population for MEDI7510: All participants in the ATP who had no major protocol deviations judged to have the potential to interfere with the generation or interpretation of an immune response to MEDI7510.
Measure: Geometric Mean (95% Confidence Interval); unit: Fragment antigen-binding (F AB) unit/mL
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 947 | 946
Fragment antigen-binding (F AB) unit/mL
  Day 1: number analyzed (Participants) | 944 | 940
  Day 1 | 83.39 [78.91 to 88.12] | 77.96 [73.66 to 82.50]
  Day 29: number analyzed (Participants) | 926 | 924
  Day 29 | 80.05 [75.68 to 84.68] | 999.03 [944.40 to 1056.81]
  End of Season 1: number analyzed (Participants) | 852 | 857
  End of Season 1 | 79.95 [75.27 to 84.93] | 370.88 [350.90 to 391.99]

4. Secondary Outcome: Geometric Mean Fold Change of Serum Antibodies Concentration Against RSV by Anti-F IgG Assay
Description: Anti-F IgG antibodies concentration was determined by a multiplex IgG assay developed on the Meso Scale discovery platform. It was calculated as: anti-log2 [mean (log2 yi)], where "yi" is the post dose antibody concentration or T-cell count fold change from baseline for each participant. The Season 1 was approximately 1 year.
Time Frame: Day 29 and End of Season 1 (approximately 1 year)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 947 | 946
Fold Change
  Day 29: number analyzed (Participants) | 926 | 924
  Day 29 | 0.96 [0.94 to 0.98] | 12.78 [11.96 to 13.65]
  End of Season 1: number analyzed (Participants) | 852 | 857
  End of Season 1 | 0.94 [0.91 to 0.96] | 4.60 [4.34 to 4.88]

5. Secondary Outcome: Percentage of Participants Who Had a Post-dose Seroresponse to RSV as Measured by Anti-F IgG Assay
Description: Anti-F IgG antibodies were determined by a multiplex IgG assay developed on the Meso Scale discovery platform. Seroresponse was defined as a greater than or equal to (>=) 3-fold rise of serum antibodies against RSV from baseline. The Season 1 was approximately 1 year.
Time Frame: Day 29 and End of Season 1 (approximately 1 year)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 947 | 946
Percentage of Participants
  Day 29: number analyzed (Participants) | 926 | 924
  Day 29 | 0.8 [0.3 to 1.5] | 92.9 [91 to 94.4]
  End of Season 1: number analyzed (Participants) | 852 | 857
  End of Season 1 | 1.6 [0.9 to 2.7] | 65.8 [62.5 to 69]

6. Secondary Outcome: Geometric Mean Titers (GMTs) of Strain-Specific Hemagglutination Inhibition (HAI) Antibodies to Influenza Antigens Contained in the Seasonal Influenza Vaccine
Description: GMT was calculated as: anti-log2 [mean (log2 xi)], where "xi" is an antibodies concentration of participants. GMTs of strain-Specific HAI antibodies (H1N1, H3N2, B Brisbane, and B Phuket) were reported. The Season 1 was approximately 1 year.
Time Frame: Day 1 (post-dose) and Day 29 of Season 1
Population: Immunogenicity population for IIV: All participants in the ATP who had no major protocol deviations judged to have the potential to interfere with the generation or interpretation of an immune response to the influenza vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 464 | 451
Titer
  H1N1, Day 1: number analyzed (Participants) | 462 | 450
  H1N1, Day 1 | 54.26 [48.610 to 60.565] | 55.77 [50.066 to 62.115]
  H1N1, Day 29: number analyzed (Participants) | 460 | 450
  H1N1, Day 29 | 161.26 [146.241 to 177.823] | 155.14 [141.356 to 170.264]
  H3N2, Day 1: number analyzed (Participants) | 462 | 450
  H3N2, Day 1 | 34.81 [31.224 to 38.804] | 35.99 [32.271 to 40.136]
  H3N2, Day 29: number analyzed (Participants) | 460 | 450
  H3N2, Day 29 | 291.73 [260.581 to 326.604] | 269.58 [241.784 to 300.569]
  B BRISBANE, Day 1: number analyzed (Participants) | 462 | 450
  B BRISBANE, Day 1 | 12.89 [11.851 to 14.025] | 13.46 [12.357 to 14.672]
  B BRISBANE, Day 29: number analyzed (Participants) | 460 | 450
  B BRISBANE, Day 29 | 32.49 [29.314 to 36.007] | 30.15 [27.334 to 33.257]
  B PHUKET, Day 1: number analyzed (Participants) | 462 | 450
  B PHUKET, Day 1 | 11.42 [10.514 to 12.402] | 11.81 [10.857 to 12.841]
  B PHUKET, Day 29: number analyzed (Participants) | 460 | 450
  B PHUKET, Day 29 | 30.00 [27.088 to 33.219] | 28.29 [25.526 to 31.348]

7. Secondary Outcome: Post-dose Geometric Mean Fold Change of Strain-Specific HAI Antibodies to Influenza Antigens Contained in the Seasonal Influenza Vaccine
Description: Geometric mean fold change was calculated as: anti-log2 [mean (log2 yi)], where "yi" is the post dose antibody concentration or T-cell count fold change from baseline for each participant. Geometric mean fold change of strain-specific HAI antibodies (H1N1, H3N2, B BRISBANE, and B PHUKET) were reported. The Season 1 was approximately 1 year.
Time Frame: Day 29 of Season 1
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 464 | 451
Fold Change
  H1N1: number analyzed (Participants) | 460 | 450
  H1N1 | 2.97 [2.652 to 3.329] | 2.78 [2.501 to 3.094]
  H3N2: number analyzed (Participants) | 460 | 450
  H3N2 | 8.42 [7.525 to 9.421] | 7.49 [6.669 to 8.414]
  B BRISBANE: number analyzed (Participants) | 460 | 450
  B BRISBANE | 2.53 [2.301 to 2.771] | 2.24 [2.068 to 2.425]
  B PHUKET: number analyzed (Participants) | 460 | 450
  B PHUKET | 2.63 [2.419 to 2.850] | 2.40 [2.217 to 2.589]

8. Secondary Outcome: Percentage of Participants Who Had a Strain-specific Post-dose Seroresponse to HAI Antibody
Description: Seroresponse was defined as a >= 4-fold rise of strain-specific HAI antibodies (H1N1, H3N2, B BRISBANE, and B PHUKET) from baseline. The Season 1 was approximately 1 year.
Time Frame: Day 29 of Season 1
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 464 | 451
Percentage of Participants
  H1N1: number analyzed (Participants) | 460 | 450
  H1N1 | 32.6 | 32.4
  H3N2: number analyzed (Participants) | 460 | 450
  H3N2 | 76.5 | 74.2
  B BRISBANE: number analyzed (Participants) | 460 | 450
  B BRISBANE | 31.7 | 26.9
  B PHUKET: number analyzed (Participants) | 460 | 450
  B PHUKET | 33.0 | 30.2

9. Secondary Outcome: Post-dose GMTs of Serum Antibodies Against RSV by Microneutralization Assay
Description: Microneutralization assay was to be used to assess humoral immunity (HAI antibody titers) against RSV. GMT was to be calculated as: anti-log2 [mean (log2 xi)], where "xi" is an antibodies concentration of participants. The Season 1 was approximately 1 year.
Time Frame: Day 29 and End of Season 1 (approximately 1 year)
Population: Data for this outcome measure were not collected as the study was terminated prematurely because the study did not meet its primary efficacy outcome measure.
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Post-dose Geometric Mean Fold Change of Serum Antibodies Against RSV by Microneutralization Assay
Description: Microneutralization assay was to be used to assess humoral immunity (HAI antibody titers) against RSV. Geometric mean fold change was to be calculated as: anti-log2 [mean (log2 yi)], where "yi" is the post dose antibody concentration or T-cell count fold rise from baseline for each participant. The Season 1 was approximately 1 year.
Time Frame: Day 29 and End of Season 1 (approximately 1 year)
Population: as for outcome 9
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Percentage of Participants Who Had a Post-dose Seroresponse to RSV by Microneutralization Assay
Description: Microneutralization assay was to be used to assess humoral immunity (HAI antibody titers) against RSV. Seroresponse was defined as a >= 3-fold rise of Serum Antibodies against RSV from baseline. The Season 1 was approximately 1 year.
Time Frame: Day 29 and End of Season 1 (approximately 1 year)
Population: as for outcome 9
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Post-dose Geometric Mean Concentration (GMC) of Palivizumab Competitive Antibodies as Measured by a Palivizumab Competitive Enzyme Linked Immunosorbent Assay (cELISA)
Description: Palivizumab cELISA assay was to be used to assess humoral immunity (HAI antibody titers) against RSV. GMC was to be calculated as: anti-log2 [mean (log2 xi)], where "xi" is an antibodies concentration of participants. The Season 1 was approximately 1 year.
Time Frame: Day 29 and End of Season 1 (approximately 1 year)
Population: as for outcome 9
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Post-dose Geometric Mean Fold Change of Palivizumab Competitive Antibodies as Measured by a Palivizumab cELISA
Description: Palivizumab cELISA assay was to be used to assess humoral immunity (HAI antibody titers) against RSV. Geometric mean fold change was to be calculated as: anti-log2 [mean (log2 yi)], where "yi" is the post dose antibody concentration or T-cell count fold rise from baseline for each participant. The Season 1 was approximately 1 year.
Time Frame: Day 29 and End of Season 1 (approximately 1 year)
Population: as for outcome 9
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Percentage of Participants Who Had a Post-dose Seroresponse to RSV as Measured by a Palivizumab cELISA
Description: Palivizumab cELISA assay was to be used to assess humoral immunity (HAI antibody titers) against RSV. Seroresponse was defined as a >= 3-fold rise of Serum Antibodies against RSV from baseline. The Season 1 was approximately 1 year.
Time Frame: Day 29 and End of Season 1 (approximately 1 year)
Population: as for outcome 9
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Participants With Any Solicited Symptoms
Description: Solicited symptoms: tenderness or soreness at site of injection, pain at site of injection, fatigue or tiredness, headache, generalized muscle aches, swelling at the site of injection, redness at the site of injection, fever >= 100.4 degrees Fahrenheit by any route from Day 1 to Day 7.
Time Frame: Day 1 (post-dose) through Day 7
Population: ATP: Participants who received any dose of investigational product (IP). Participants were included in the ATP according to the IP received even if different from that to which the participant was randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 948 | 946
Participants | 558 | 606

16. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent events were between administration of study drug and Day 29 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Day 1 (post-dose) through Day 29
Population: ATP: Participants who received any dose of IP. Participants were included in the ATP according to the IP received even if different from that to which the participant was randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 948 | 946
Participants | 141 | 146

17. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events of Special Interest (TEAESIs), Treatment-Emergent Serious Adverse Events (TESAEs) and Treatment-Emergent New Onset Chronic Disease (NOCDs)
Description: An serious adverse event (SAE) was an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between administration of study drug and approximately 1 year follow up that were absent before treatment or that worsened relative to pretreatment state. An adverse event of special interest was one of scientific and medical interest specific to understanding of study drug and may have required close monitoring and rapid communication by investigator to the sponsor. A NOCD was a newly diagnosed medical condition that is of a chronic, ongoing nature. It was observed after receiving study drug and was assessed by investigator as medically significant. The Season 1 was approximately 1 year.
Time Frame: Day 1 (post-dose) through end of Season 1 (approximately 1 year)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + IIV | MEDI7510 + IIV
Number analyzed (Participants) | 948 | 946
Participants
  TEAESIs | 0 | 1
  TESAEs | 3 | 4
  NOCDs | 5 | 4

ADVERSE EVENTS:
Time Frame: Day 1 (post-dose) through end of Season 1 (approximately 1 year)
Groups:
- MEDI7510+IIV: Participants received a single IM injection of MEDI7510 in one arm and single IM injection of IIV in the contralateral arm.
Arm/Group | Placebo + IIV | MEDI7510+IIV
All-Cause Mortality (participants affected / at risk) | 5/948 | 3/946
Serious Adverse Events (participants affected / at risk) | 57/948 | 64/946
Other Adverse Events (participants affected / at risk) | 52/948 | 48/946
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + IIV (N=948) | MEDI7510+IIV (N=946)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2) | 2 (2)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 4 (5)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 6 (7) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis relapsing (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Infected lymphocele (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Device failure (Product Issues) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Drug dependence (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic occlusion (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + IIV (N=948) | MEDI7510+IIV (N=946)
Fatigue (General disorders) | 11 (13) | 16 (19)
Injection site pain (General disorders) | 18 (35) | 10 (28)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 16 (16)
Viral upper respiratory tract infection (Infections and infestations) | 10 (10) | 13 (13)
Headache (Nervous system disorders) | 13 (15) | 10 (11)

LIMITATIONS AND CAVEATS:
The study was terminated due to failure to meet the primary efficacy endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.